CLINICAL TRIAL: NCT04247672
Title: The ATtune Knee Outcome Study: Prospective Evaluation of a Novel Uncemented Rotating Platform Total Knee Arthroplasty
Brief Title: The ATtune Knee Outcome Study
Acronym: ATKOS
Status: Recruiting | Type: Observational
Sponsor: Spaarne Gasthuis (Other)
Responsible Party: Sponsor
Other Study IDs: 2019.0084
Record Dates: First submitted 2020-01-20; First posted 2020-01-30 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Osteoarthritis, Knee; Knee Osteoarthritis; Knee Rheumatism; Rheumatoid Arthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Arthritis, Rheumatoid | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Total Knee Arthroplasty (uncemented rotating platform ATTUNE) — All patients receive an uncemented ATTUNE rotating platform knee system.
  Other Names: Total knee arthroplasty

SUMMARY:
To accomodate dissatisfied patients with a total knee arthroplasty (TKA) and improve outcomes, several knee systems have been developed. The cemented ATTUNE TKA shows superiority over other established knee systems at short-term, abating with longer follow-up. There have been no studies reporting on the results of the uncemented version of the ATTUNE. Therefore, the main objective of the current study was to report patient reported outcome measures (PROMs), survivorship and complications associated with the uncemented ATTUNE TKA.

DETAILED DESCRIPTION:
Every year, 1.5 million total knee arthroplasties (TKA) are performed worldwide in patients whose joints have been severely affected by osteoarthritis, rheumatoid arthritis, or trauma, causing intense pain and loss of function. Due to the ageing society, these numbers are expected to have increased six-fold to 3.48 million cases annually by 2030. Even though joint replacement provides satisfactory and durable results for most patients, 20% is thought to still not be satisfied with their artificial joint. To accommodate this dissatisfied population and improve durability of implants even more, several knee systems have been developed over the years. One of the newest models is the ATTUNE knee system (DePuy, Warsaw, Indiana, USA). One of the landmark features is a gradually reducing radius in the geometry of the femoral component, more closely mimicking the anatomical patellofemoral joint and facilitating more natural femoral rollback during flexion. Comparisons of the cemented ATTUNE with previous knee systems show promising results in terms of patellofemoral outcomes, but fail to demonstrate definitive superiority in terms of all patient reported outcomes. Clinical superiority of the ATTUNE tends to abate with longer follow-up, implicating a possible superiority in the short-term recovery and return to activities. There is no follow-up study reporting the results of the uncemented ATTUNE. Moreover, all previously cited studies report better patellofemoral outcomes with patellar resurfacing, making it still unclear whether the implicated superior design changes of the femoral component hold ground without patellar resurfacing.

The primary objective is to report survivorship, complications and patient reported outcome measures associated with the uncemented ATTUNE rotating platform knee system. Secondary objectives are (1) evaluate patient reported (patellofemoral) outcomes (2) assess return to work and sport after TKA (3) translate and validate the Dutch version of the University of California, Los Angeles (UCLA) activity scale and (4) analyse psychologic factors (such as pain catastrophising and coping) and the impact on dissatisfaction following TKA.

ELIGIBILITY:
Inclusion Criteria:

* End-stage osteoarthritis of the knee warranting joint replacement therapy.
* Indicated for an ATTUNE total knee system as part of regular clinical practice.
* Capability and willingness to sign informed consent and comply with follow-up procedures.
* Capable enough in Dutch or English to be able to understand study procedures

Exclusion Criteria:

* Unable or unwilling to sign informed consent and comply with follow-up
* Indication for primary revision arthroplasty
* Absolute indication for cemented fixation (decreased bone stock/quality of spongiosa)

Ages: 21 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients with end-stage knee disease (e.g. knee osteoarthritis) warranting and able to undergo knee replacement therapy.
Sampling Method: Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2020-02-03 (Actual); Primary Completion 2024-01-22 (Estimated); Study Completion 2036-01-22 (Estimated)

PRIMARY OUTCOMES:
Survivorship | 10 year
  Calculated by determining revision rate. Septic, aseptic and all-cause revision rates will be calculated seperately.
Complication rate | 10 year
  All substantial complications associated with total knee arthroplasty will be registered and reported
Forgotten Joint Score 12 (FJS-12) | 10 year
Kujala Anterior Knee Pain Scale (AKPS) | 10 year
Knee injury and Osteoarthritis Outcome Scale - Physical Function Short Form | 10 year
  KOOS-PS
Numeric Rating Scale (NRS) | 10 year
  NRS on pain and satisfaction
EuroQol 5 Dimensions, 3 Levels (EQ5D-3L) | 10 year

SECONDARY OUTCOMES:
30 second chair stand test (30sCST) | 1 year
  The amount of times one can stand up and sit down from a chair in 30 seconds
40m Fast paced walk test (40m-FPWT) | 1 year
  The amount of seconds one does to walk 40 meters.
Stair climb test (SCT) | 1 year
  The time one takes to walk a set of stairs up and down.
Tegner activity rating scale | 1 year
  1-item questionnaire
University of California, Los Angeles (UCLA) activity rating scale | 1 year
  1-item questionnaire
Return to work | 1 year
  Assessed by a short self-composed questionnaire, which evaluates what kind of work the patients do, when they started after surgery and whether this is the same as their preoperative job
Alignment | 1 year
  A long-leg radiograph is performed 1 year after surgery to assess mechanical alignment of the prosthesis with consideration of femur and tibia
Patient Health Questionnaire (PHQ-2) | 10 year
  2-item questionnaire to screen for major depressive episodes
Pain Self Efficacy Questionnaire (PSEQ) | 10 year
  Questionnaire to asses pain self efficacy
Pain Catastrophizing Scale (PCS) | 10 year
  Explores pain catastrophizing and its relation to pain behaviour

CONTACTS AND LOCATIONS:
Locations (1):
- Spaarne Gasthuis, Hoofddorp, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rassir R, Sierevelt IN, Schager M, Nolte PA; ATKOS group. Design and rationale of the ATtune Knee Outcome Study (ATKOS): multicenter prospective evaluation of a novel uncemented rotating platform knee system. BMC Musculoskelet Disord. 2021 Jul 15;22(1):622. doi: 10.1186/s12891-021-04493-1. PMID 34266444